CLINICAL TRIAL: NCT06953232
Title: Acute Impact of Whey Protein-enriched Milk Fat Globule Membrane Supplementation on Postprandial Markers of Heart and Brain Health in Postmenopausal Women Living With Overweight and at Moderate Risk for Cardiovascular Disease.
Brief Title: Acute Impact of Whey Protein-enriched Milk Fat Globule Membrane Supplementation on Postprandial Markers of Heart and Brain Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Dr Oonagh Markey, Principal Investigator, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Project ID: 18721
Record Dates: First submitted 2025-04-15; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Diseases; Cognition; Overweight or Obesity; Postmenopausal Women; Cardiometabolic Risk Factors
Keywords: Milk fat globule membrane; Milk polar lipids; triacylglycerol; postprandial; cholesterol; cardiometabolic disease risk; cognitive function
MeSH Terms: conditions — Cardiovascular Diseases; Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to the assignment of intervention or control. Data analysis will be conducted in a blinded manner to reduce potential bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whey protein-enriched milk fat globule membrane supplement (Experimental): Participants will consume a high-fat, mixed meal containing approximately 75 g of test fat (refined palm oil), supplemented with a whey protein-enriched milk fat globule membrane (providing ~5 g of milk polar lipids) powdered ingredient. The experimental and placebo meals will be isoenergetic and protein-matched, and will be administered in a randomised order, with a washout period of at least 21 days between sessions.
  Interventions: Dietary Supplement: Whey protein-enriched milk fat globule membrane supplement
- Whey protein-based supplement (Placebo Comparator): Participants will consume a high-fat, mixed meal containing approximately 75 g of test fat (refined palm oil) supplemented with a whey protein-based powdered ingredient without milk fat globule membrane (placebo) The experimental and placebo meals will be isoenergetic and protein-matched, and will be administered in a randomised order, with a washout period of at least 21 days between sessions.
  Interventions: Dietary Supplement: Whey protein-based supplement

INTERVENTIONS:
Dietary Supplement: Whey protein-enriched milk fat globule membrane supplement — Participants will consume a high-fat, mixed meal containing approximately 75 g of test fat (refined palm oil), supplemented with a whey protein-enriched milk fat globule membrane (providing ~5 g of milk polar lipids) powdered ingredient. The experimental and placebo meals will be isoenergetic and protein-matched, and will be administered in a randomised order, with a washout period of at least 21 days between sessions.
  Arms: Whey protein-enriched milk fat globule membrane supplement
Dietary Supplement: Whey protein-based supplement — Participants will consume a high-fat, mixed meal containing approximately 75 g of test fat (refined palm oil) supplemented with a whey protein-based powdered ingredient without milk fat globule membrane (placebo) The experimental and placebo meals will be isoenergetic and protein-matched, and will be administered in a randomised order, with a washout period of at least 21 days between sessions.
  Other Names: Placebo
  Arms: Whey protein-based supplement

SUMMARY:
In a single-blind, randomised, placebo-controlled crossover manner, this study aims to assess the impact of a high-fat mixed meal containing a whey protein (WP)-enriched milk fat globule membrane (MFGM) powdered ingredient on markers of heart and brain health in the fed state among middle-to-older-aged, postmenopausal women living with overweight and at moderate risk for cardiovascular disease.

Participants will attend two ~8 hour study visits, where they will consume a high-fat meal containing a WP-enriched MFGM powdered ingredient or a placebo WP-based powdered ingredient. Each visit will involve anthropometric measurements and periodic assessments of heart health, including blood pressure and blood vessel stiffness measurements, blood sample collections, as well as computer-based tests measuring mood and cognition (brain function) over a 6-hour postprandial period.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy postmenopausal women (not menstruating for 12 or more months)
* Aged 50 - 70 years
* BMI: 25 - 40 kg/m²
* Moderate CVD risk
* Recreationally active (> 3 x 30 min moderate exercise per week)
* Understands and is willing and able to comply with all study procedures including eating a high-fat breakfast meal
* Fluent in written and spoken English
* Access to, and able to use, the internet/computer/tablet device

Exclusion Criteria:

* Smoking (including vaping)
* Diagnosed with cardiovascular disease or suffered myocardial infarction /stroke in the past twelve months
* Existing or significant past medical history of any medical condition likely to affect the study outcomes e.g., diabetes, digestive, cancer or thyroidal disease, neurological disease (Alzheimer's disease, other form of dementia, mild cognitive impairment), or serious mental illness know to affect cognition (schizophrenia, schizoaffective disorder, bipolar disorder), learning disorders (dyslexia)
* Early or premature menopause resulting from medical conditions or undergoing surgery
* Hormone replacement therapy within last 6 months
* Prescribed medications likely to interfere with study outcomes (including lipid/cholesterol-lowering medications, including statins; blood thinners, antiplatelets (anticoagulants) such as heparin, etc.; medications for blood pressure; inflammation such as nonsteroidal anti-inflammatory drugs, aspirin, etc.; immune function, or lipid/carbohydrate metabolism) or prescribed antibiotics within the last three months
* Use of antidepressant or anti-anxiety medication if it has changed in the last three months or expected to change within the 3-month study period
* Taking vitamin, mineral, or fatty acid supplements (e.g., fish oil, calcium) or unwilling stop consuming these for the duration of the study (including sufficient washout period)
* Working night shifts
* Inaccessible veins for blood collection via cannulation
* Unstable weight history (≥3 kg loss or gain in the previous 3 months) or planning or currently on a weight reduction scheme
* Known allergy or intolerance to study food (including lactose intolerance, dairy, and wheat)
* Being vegan or any other unusual medical history or diet and lifestyle habits or practices that would preclude volunteers from participating in a dietary intervention or metabolic study
* Excessive alcohol consumption: >21 unit/wk (i.e., more than 10 and a half pints of beer or 21 small glasses of wine)
* Currently taking part or have participated in another research study in the last two months (e.g., dietary intervention)

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Postprandial change in circulating triacylglycerol response, assessed by iAUC 0-360 min. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Measured using a spectrophotometric assay or high-throughput 1H-NMR metabolomics platform.

SECONDARY OUTCOMES:
Postprandial change in circulating triacylglycerol response, assessed via AUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Measured using a spectrophotometric assay or high-throughput 1H-NMR metabolomics platform.
Postprandial change in circulating triacylglycerol response, assessed via Cₘₐₓ. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Measured using a spectrophotometric assay or high-throughput 1H-NMR metabolomics platform.
Postprandial change in circulating triacylglycerol response, assessed via Tₘₐₓ. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Measured using a spectrophotometric assay or high-throughput 1H-NMR metabolomics platform.
Postprandial change in circulating triacylglycerol response, assessed via time-course profile. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Measured using a spectrophotometric assay or high-throughput 1H-NMR metabolomics platform.
Postprandial change in circulating lipid and apolipoprotein responses, assessed via AUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Measured using a spectrophotometric assay or high-throughput 1H-NMR metabolomics platform.
Postprandial change in circulating lipid and apolipoprotein responses, assessed via iAUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Measured using a spectrophotometric assay or high-throughput 1H-NMR metabolomics platform.
Postprandial change in circulating lipid and apolipoprotein responses, assessed via Cₘₐₓ. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Measured using a spectrophotometric assay or high-throughput 1H-NMR metabolomics platform.
Postprandial change in circulating lipid and apolipoprotein responses, assessed via Tₘₐₓ. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Measured using a spectrophotometric assay or high-throughput 1H-NMR metabolomics platform.
Postprandial change in circulating lipid and apolipoprotein responses, assessed via time-course profiles. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Measured using a spectrophotometric assay or high-throughput 1H-NMR metabolomics platform.
Postprandial changes in circulating lipoprotein subclass particle size and concentrations, assessed via AUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Assessed using high-throughput 1H-NMR metabolomics platform.
Postprandial changes in circulating lipoprotein subclass particle size and concentrations, assessed via iAUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Assessed using high-throughput 1H-NMR metabolomics platform.
Postprandial changes in circulating lipoprotein subclass particle size and concentrations, assessed via Cₘₐₓ. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Assessed using high-throughput 1H-NMR metabolomics platform.
Postprandial changes in circulating lipoprotein subclass particle size and concentrations, assessed via Tₘₐₓ. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Assessed using high-throughput 1H-NMR metabolomics platform.
Postprandial changes in circulating lipoprotein subclass particle size and concentrations, assessed via time-course profiles. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Assessed using high-throughput 1H-NMR metabolomics platform.
Postprandial change in circulating apolipoprotein B48 response, assessed via AUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by ELISA.
Postprandial change in circulating apolipoprotein B48 response, assessed via iAUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by ELISA.
Postprandial change in circulating apolipoprotein B48 response, assessed via time-course profile. | Blood samples will be taken at -60, 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by ELISA.
Postprandial change in circulating glucose response, assessed via AUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Measured using a spectrophotometric assay or high-throughput 1H-NMR metabolomics platform.
Postprandial change in circulating glucose response, assessed via iAUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Measured using a spectrophotometric assay or high-throughput 1H-NMR metabolomics platform.
Postprandial change in circulating glucose response, assessed via Cₘₐₓ. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Measured using a spectrophotometric assay or high-throughput 1H-NMR metabolomics platform.
Postprandial change in circulating glucose response, assessed via Tₘₐₓ. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Measured using a spectrophotometric assay or high-throughput 1H-NMR metabolomics platform.
Postprandial change in circulating glucose response, assessed via timecourse profile. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Measured using a spectrophotometric assay or high-throughput 1H-NMR metabolomics platform.
Postprandial change in circulating insulin response, assessed via AUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Determined by ELISA.
Postprandial change in circulating insulin response, assessed via iAUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Determined by ELISA.
Postprandial change in circulating insulin response, assessed via Cₘₐₓ. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Determined by ELISA.
Postprandial change in circulating insulin response, assessed via Tₘₐₓ. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Determined by ELISA.
Postprandial change in circulating insulin response, assessed via timecourse profile. | Blood samples will be taken at -60, 0 (baseline) and 30, 60, 90, 120, 180, 240, 300, 360 minutes (after meal ingestion)
  Determined by ELISA.
Postprandial change in circulating interleukin-6 response, assessed via AUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by ELISA
Postprandial change in circulating interleukin-6 response, assessed via iAUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by ELISA
Postprandial change in circulating interleukin-6 response, assessed via time-course profile. | Blood samples will be taken at -60, 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by ELISA
Postprandial change in circulating soluble CD14 response, assessed via AUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by ELISA
Postprandial change in circulating soluble CD14 response, assessed via iAUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by ELISA
Postprandial change in circulating soluble CD14 response, assessed via time-course profile. | Blood samples will be taken at -60, 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by ELISA
Postprandial change in circulating lipopolysaccharide-binding protein response, assessed via AUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by ELISA
Postprandial change in circulating lipopolysaccharide-binding protein response, assessed via iAUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by ELISA
Postprandial change in circulating lipopolysaccharide-binding protein response, assessed via time-course profile. | Blood samples will be taken at -60, 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by ELISA
Postprandial change in responses of selected circulating gut-related metabolite (for example, trimethylamine N-oxide, and short-chain fatty acids), assessed via AUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by ELISA
Postprandial change in responses of selected circulating gut-related metabolite (for example, trimethylamine N-oxide, and short-chain fatty acids), assessed via iAUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by ELISA
Postprandial change in responses of selected circulating gut-related metabolite (for example, trimethylamine N-oxide, and short-chain fatty acids), assessed via time-course profiles. | Blood samples will be taken at -60, 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by ELISA
Postprandial change in clinic systolic and diastolic blood pressure, assessed via AUC₀-₃₆₀min. | Measurements will be taken at 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by automated upper arm sphygmomanometer
Postprandial change in clinic systolic and diastolic blood pressure, assessed via iAUC₀-₃₆₀min. | Measurements will be taken at 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by automated upper arm sphygmomanometer
Postprandial change in clinic systolic and diastolic blood pressure, assessed via time-course profiles. | Measurements will be taken at 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by automated upper arm sphygmomanometer
Postprandial change in markers of arterial stiffness including augmentation index and augmentation index adjusted to a standard heart rate of 75 bpm, assessed via AUC₀-₃₆₀min. | Measurements will be taken at 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by radial pulse wave analysis (using applanation tonometry)
Postprandial change in markers of arterial stiffness including augmentation index and augmentation index adjusted to a standard heart rate of 75 bpm, assessed via iAUC₀-₃₆₀min. | Measurements will be taken at 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by radial pulse wave analysis (using applanation tonometry)
Postprandial change in markers of arterial stiffness including augmentation index and augmentation index adjusted to a standard heart rate of 75 bpm, assessed via time-course profiles. | Measurements will be taken at 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by radial pulse wave analysis (using applanation tonometry)
Postprandial change in cognitive test performance. | Test battery will be completed at 0 (baseline) and 240 minutes (after meal ingestion)
  Cognition will be assessed using a neuropsychological nine-test battery which assesses global and domain-specific function, as determined by NeurOn software.
Postprandial change in mood. | Questionnaire will be completed at 0 (baseline) and 240 minutes (after meal ingestion)
  Determined by the Bond-Lader visual analogue scale (includes 16 items each having antonyms on two ends, on a scale of 1 to 100, 50 being the neutral point)
Postprandial change in responses of selected circulating biomarkers of cognitive health/neuroinflammation (for example, brain-derived neurotrophic factor), assessed via AUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by ELISA
Postprandial change in responses of selected circulating biomarkers of cognitive health/neuroinflammation (for example, brain-derived neurotrophic factor), assessed via iAUC₀-₃₆₀min. | Blood samples will be taken at -60, 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by ELISA
Postprandial change in responses of selected circulating biomarkers of cognitive health/neuroinflammation (for example, brain-derived neurotrophic factor), assessed via time-course profiles. | Blood samples will be taken at -60, 0 (baseline) and 120, 240, 360 minutes (after meal ingestion)
  Determined by ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No